CLINICAL TRIAL: NCT04215393
Title: An Exploratory Clinical Trial Evaluating the Tolerability and Efficacy of Conbercept Eye Drops in Patients With Corneal Neovascularization
Brief Title: An Exploratory Clinical Trial Evaluating the Tolerability and Efficacy of KH906 in Patients With Corneal Neovascularization
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: KH906-40101
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conbercept eye drop (0.1mg/ mL) (Experimental): Subjects in this arm will receive 0.1mg/mL Conbercept eye drop 4 times a day, one drop at a time.
  Interventions: Drug: Conbercept eye drop
- Conbercept eye drop (0.5mg/ mL) (Experimental): Subjects in this arm will receive 0.5mg/mL Conbercept eye drop 4 times a day, one drop at a time.
  Interventions: Drug: Conbercept eye drop; Drug: Placebo
- Conbercept eye drop (1.0mg/ mL) (Experimental): Subjects in this arm will receive 1.0mg/mL Conbercept eye drop 4 times a day, one drop at a time.
  Interventions: Drug: Conbercept eye drop; Drug: Placebo

INTERVENTIONS:
Drug: Conbercept eye drop — In the first stage, subjects will be receive Conbercept eye drop. In the second stage,subjests will revceive conbercept eye drop or placebo.
Drug: Placebo — In the second stage, subjects will be receive Conbercept eys drop or a placebo.
  Arms: Conbercept eye drop (0.5mg/ mL); Conbercept eye drop (1.0mg/ mL)

SUMMARY:
The first stage of this study will evaluates the tolerability of different concentrations of Conbercept eye drop to patients with corneal neovascularization.

The second stage of this study will evaluate the effectiveness of conbercept eye drop initially.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form, volunteered to participate in the trial and followed up according to the protocol.
* Ages from 18 to 75,male or female.
* Superficial or deep neovascularization induced by trauma/chemical burn/inflammation/corneal transplantation.

Exclusion Criteria:

* Subjects who had significant defect in the corneal epithelium.
* Study eye had been injected of anti-vegf drugs within 3 months before screening
* Study eye was performed surgery (except keratoplasty) within 3 months prior screening, or eye surgery was planned during this trial period.
* Oral glucocorticoid administration within 1 month prior screening (except for duration less than 7 days)
* Systemic use of anti-vegf drugs within 45 days prior to screening.
* Have history of abnormal coagulation, such as end-stage liver disease, or are taking anticoagulants（except aspirin）.
* Uncontrolled clinical problems such as canner etc..
* Unable or unwilling to use effective contraception.
* Positive blood tests for pregnancy (female subjects)
* Participated in drug clinical trials within 3 months before the first administration.
* The researchers think the participants were not suitable for this trail.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Ocular and Systemic Safety: occurrence of ocular and systemic adverse events | day 14
  The occurrence of ocular and systemic adverse events was closely monitored over the course of this study. Ocular adverse events were monitored through complete ocular examinations. Systemic adverse events were identified with physical examinations.

SECONDARY OUTCOMES:
The Size and Extent of Corneal Neovascularization Will be Measured by Computerized Image Analysis of Corneal Photographs Taken Throughout the Study | day 14 and day 28
  The efficacy of KH906 in the treatment of corneal NV was evaluated by comparing corneal photographs taken at baseline with corneal photographs taken at the follow-up visits. Percent change from baseline was measured.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No